CLINICAL TRIAL: NCT02283567
Title: The Difference Between Elasticity of the Uterine Cervix in Singleton and Twin Pregnancies
Acronym: DEU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Rami Aviram, MD, Meir Medical Center
Other Study IDs: 0152-14-MMC
Record Dates: First submitted 2014-10-27; First posted 2014-11-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators aim to compare elasticity of the uterine cervix in singleton and twin pregnancies of similar gestational age.

DETAILED DESCRIPTION:
Softening of the uterine cervix occurs during pregnancy.There is a possibility that this process occurs earlier in twin versus singleton pregnancies.The softening of the cervix is reflected by the level of its elasticity which can be measured sonoelastographically. A two dimension image of the cervix is obtained in the midsagittal section and the length is noted. A 2nd sonoelastography image is obtained before pressure is applied with the transducer in the area of the internal os and a third sonoelastography image is obtained until no more shortening of the anterior-posterior diameter is observed.Elastography measurements of the internal os are performed using a color map: red (soft), yellow (medium soft), blue (medium hard) and purple (hard) before and after the application of strain.The change between the color maps before and after strain application in singleton pregnancies will be compared to the change in twin pregnancies of similar gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Low risk singleton and twin pregnancies

Exclusion Criteria:

* Patients with pregnancy complications

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20-44 years old pregnant patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of elasticity levels in singleton and twin pregnancies (Elastographic measurements of the internal os) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rami Aviram, MD, Principal Investigator — Meir Medical Center